CLINICAL TRIAL: NCT06293053
Title: A Multicenter Open-label Study to Investigate the Pharmacokinetics and Safety of Dupilumab in Participants ≥6 Months to <18 Years of Age With Prurigo Nodularis
Brief Title: A Study to Investigate the Pharmacokinetics and Safety of Dupilumab in Participants ≥6 Months to <18 Years of Age With Prurigo Nodularis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKM17836; U1111-1287-7255 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Prurigo Nodularis
MeSH Terms: interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dupilumab (Experimental): Administered subcutaneously (SC) based on weight and age
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — Pharmaceutical form: Injection solution
  Route of administration: Subcutaneous
  Other Names: SAR231893; Dupixent

SUMMARY:
This is a Phase 3, multicenter, open-label, pharmacokinetics (PK)/safety study.

The study consists of 3 periods:

* Screening period: 2 to 4 weeks.
* Treatment period: 24 weeks.
* Post-intervention follow-up period: 16 weeks. The study duration will be approximately 42 to 44 weeks for each participant (including screening, treatment, and follow-up periods).

The total number of planned study visits for each participant will be 6.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥6 months to <18 years of age, at the time of signing the informed consent.
* A clinical diagnosis of prurigo nodularis (PN) at least 3 months prior to screening, an Investigator's global assessment for prurigo nodularis stage (IGA PN-S) score of ≥2 with presence of ≥6 pruriginous lesions at Baseline. The lesions should be present on ≥2 different body surface areas at Baseline.
* On the worst itch numerical rating scale (WI-NRS) (for participants aged ≥6 years to <18 years old at the screening visit) or worst-scratch/itch NRS (for participants aged ≥6 months to <6 years at the screening visit) ranging from 0 to 10, participants must have an average worst itch score of ≥7 in the 7 days prior to Day 1.

NOTE: Baseline pruritus NRS average score for maximum itch intensity will be determined based on the average of daily NRS scores for maximum intensity (the daily score ranges from 0 to 10) during the 7 days immediately preceding the Day 1/Baseline visit. A minimum of 4 daily scores out of the 7 days is required to calculate the baseline average score.

* Participants/Caregivers must be willing and able to complete a daily symptom e-Diary for the duration of the study.
* Contraceptive use by male and female participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Presence of active moderate to severe lesions of atopic dermatitis (AD), and/or other skin conditions that may interfere with the PN diagnosis including but not limited to the following: scabies, psoriasis, lymphomatoid papulosis, habitual picking, dermatitis herpetiformis, sporotrichosis, and bullous disease.
* Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, or antifungals within 2 weeks before the screening visit or during the screening period.

NOTE: Participants may be rescreened after infection resolves.

* Known or suspected immunodeficiency, including history of invasive opportunistic infections (eg, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, and aspergillosis) despite infection resolution, or otherwise recurrent infections of abnormal frequency or prolonged duration suggesting an immune compromised status, as judged by the Investigator.
* Severe concomitant illness(es) that, in the Investigator's judgment, would adversely affect the participant's participation in the study.
* Planned or anticipated major surgical procedure during the participant's participation in this clinical trial.
* Participants who has taken biologic therapy/systemic immunosuppressant/ immunomodulator within 4 weeks before the screening visit or 5 half-lives, whichever is longer.
* Current participation to any clinical trial of an investigational drug or device or participation within 3 months before the screening visit or 5 half-lives of the investigational compound, whichever is longer.
* Participation in prior dupilumab clinical study or have been treated with commercially available dupilumab.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2027-10-28 (Estimated); Study Completion 2027-11-03 (Estimated)

PRIMARY OUTCOMES:
Concentration of dupilumab in serum | Day 1 to Week 40
  Concentration of dupilumab in serum over time

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) or serious adverse events (SAEs) | Date of signed ICF (2-4 weeks before Day 1) to Week 40
Incidence of anti-drug antibodies (ADA) to dupilumab over time | Day 1 to Week 40

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Stanford University Medical Center CTRU - 800 Welch Road- Site Number : 8400021, Palo Alto, California
  - Mission Dermatology Center- Site Number : 8400011, Rancho Santa Margarita, California
  - Pediatric Center of Excellence (PCE) - Miami Pediatric Endocrinology- Site Number : 8400005, Coral Gables, Florida
  - Life Clinical Trials - Coral Springs- Site Number : 8400018, Coral Springs, Florida
  - Direct Helpers Research Center- Site Number : 8400015, Hialeah, Florida
  - SunCoast Skin Solutions - Lutz- Site Number : 8400008, Lutz, Florida
  - USF Health- Site Number : 8400003, Tampa, Florida
  - Tareen Dermatology - Eagan- Site Number : 8400022, Eagan, Minnesota
  - MediSearch Clinical Trials- Site Number : 8400004, Saint Joseph, Missouri
  - AXIS Clinicals - Fargo- Site Number : 8400013, Fargo, North Dakota
  - Vital Prospects Clinical Research Institute - Tulsa- Site Number : 8400002, Tulsa, Oklahoma
  - Dell Children's Medical Center- Site Number : 8400007, Austin, Texas
  - Driscoll Children's Hospital- Site Number : 8400017, Corpus Christi, Texas
  - Texas Dermatology and Laser Specialists - San Antonio - Oakwell Court- Site Number : 8400020, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: PKM17836 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25648&tenant=MT_SNY_9011